CLINICAL TRIAL: NCT00607997
Title: A Phase 2, Open-Label, Multicenter Clinical Study of the Safety and Efficacy of Voreloxin (Vosaroxin) Injection in Patients Equal to or Greater Than 60 Years of Age With Previously Untreated Acute Myeloid Leukemia
Brief Title: Study of Voreloxin (Vosaroxin) in Older Patients With Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunesis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPO-0014
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Leukemia; Acute Disease; Acute Myeloid Leukemia; Nonlymphocytic Leukemia; Myelodysplastic Syndromes
Keywords: Leukemia; Myeloid; Elderly; Hematologic; Blood; Cancer; Malignancy; SNS-595; Sunesis; Hematologic Diseases; Myelodysplastic Syndromes; Older; voreloxin; reveal-1
MeSH Terms: conditions — Leukemia; Acute Disease; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Neoplasms; Hematologic Diseases | interventions — vosaroxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Study Patients (Experimental): * Schedule A: 72 mg/m2 vosaroxin Days 1, 8 and 15
  * Schedule B: 72 mg/m2 vosaroxin on Days 1 and 8
  * Schedule C: 72 mg/m2 on Days 1 and 4, or
  * Schedule C: 90 mg/m2 on Days 1 and 4
  Interventions: Drug: vosaroxin

INTERVENTIONS:
Drug: vosaroxin — Vosaroxin was administered by slow intravenous (IV) infusion or via syringe pump within 10 minutes.Patients could have completed up to 4 treatment cycles consisting of 1 or 2 induction treatment cycles and up to 2 consolidation treatment cycles. For Schedule A, an induction cycle was a minimum of 21 days during which patients received vosaroxin on Days 1, 8, and 15, followed by weekly observations until hematologic recovery for patients with aplastic marrow after the postinduction bone marrow assessment. For Schedules B and C, an induction cycle was a minimum of 15 days, during which patients received vosaroxin on Days 1 and 8 (Schedule B), or Days 1 and 4 (Schedule C), followed by the same weekly observations until hematologic recovery as for Schedule A.
  Other Names: voreloxin; SNS-595

SUMMARY:
This study will evaluate the overall remission rate of treatment with vosaroxin (formerly voreloxin) Injection in patients at least 60 years of age with previously untreated AML

DETAILED DESCRIPTION:
Other objectives of this study include:

1. Assess the safety of treatment with vosaroxin, including the 30 and 60 day all-cause mortality
2. Assess leukemia free survival (LFS), event-free survival (EFS), overall survival (OS), and duration of remission (DR).
3. Characterize the pharmacokinetic (PK) profile of vosaroxin in this patient population.
4. Evaluate potential stratification biomarkers by evaluating DNA-damage and apoptotic pathways in bone marrow samples before and after treatment with vosaroxin

ELIGIBILITY:
Key Inclusion Criteria:

1. At least 60 years of age and diagnosis of previously untreated AML (either de novo or from an antecedent hematologic disorder or therapy related AML)
2. At least 20% blasts by BM biopsy or aspirate
3. ECOG performance status of 0,1,or 2
4. Adequate cardiac, renal and liver function

Key Exclusion Criteria:

1. Uncontrolled DIC
2. Active central nervous system involvement by AML
3. Requiring hemodialysis or peritoneal dialysis
4. Some prior history of heart attack or stroke (depending on how long ago the event occurred)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2008-05-15 (Actual); Primary Completion 2009-11 (Actual); Study Completion 2009-11-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Craig, MD, Study Director — Sunesis Pharmaceuticals
Locations (19):
- United States (19):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Scripps Cancer Center, La Jolla, California
  - Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado
  - Rush University Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - St. Francis Hospital & Health Systems at Beech Grove Campus, Indianapolis, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - LSU Health Sciences Center at Shreveport, Shreveport, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - University of MO Ellis Fischel Cancer Center, Columbia, Missouri
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
De-identified data of individual participants experiencing Serious Adverse Events

REFERENCES:
- [Derived] Stuart RK, Cripe LD, Maris MB, Cooper MA, Stone RM, Dakhil SR, Turturro F, Stock W, Mason J, Shami PJ, Strickland SA, Costa LJ, Borthakur G, Michelson GC, Fox JA, Leavitt RD, Ravandi F. REVEAL-1, a phase 2 dose regimen optimization study of vosaroxin in older poor-risk patients with previously untreated acute myeloid leukaemia. Br J Haematol. 2015 Mar;168(6):796-805. doi: 10.1111/bjh.13214. Epub 2014 Nov 17. PMID 25403830

RESULTS

PARTICIPANT FLOW:
Groups:
- Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15: The original Schedule A used a single arm Green Dahlberg design (Green 1992) with 30 patients planned to be treated in Stage I.
- Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8: Schedule B was to use a single arm Green Dahlberg 2 stage design with 30 patients planned to be treated in Stage I and 25 patients in Stage II.
- Schedule C: 72 mg/m2 on Days 1 and 4: Schedule C (implemented under Amendment 2) was a dosing schedule of 72 mg/m2 on Days 1 and 4, and a total of 29 patients were enrolled and treated at this dose
- Schedule C: 90 mg/m2 on Days 1 and 4: Amendment 3 added a second dose cohort to Schedule C to treat approximately 10 patients with 90 mg/m2 vosaroxin on Days 1 and 4.
Period: Overall Study
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Started | 29 | 35 | 29 | 20
Completed | 2 | 8 | 5 | 4
Not Completed | 27 | 27 | 24 | 16
Not completed — Lack of Efficacy | 6 | 20 | 14 | 10
Not completed — Death | 8 | 5 | 2 | 5
Not completed — Adverse Event | 3 | 1 | 2 | 0
Not completed — Physician Decision | 4 | 1 | 0 | 0
Not completed — Relapse, recurrent illness | 4 | 0 | 2 | 0
Not completed — Other without explanation | 2 | 0 | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Schedule C: 72 mg/m2 on Days 1 and 4: Schedule C (also implemented under Amendment 2) was a dosing schedule of 72 mg/m2 on Days 1 and 4, and a total of 29 patients were enrolled and treated at this dose
- Total: Total of all reporting groups
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4 | Total
Number analyzed (Participants) | 29 | 35 | 29 | 20 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (6.20) | 74.2 (5.85) | 70.5 (5.68) | 76.5 (5.70) | 73.6 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 15 | 3 | 40
  Male | 19 | 23 | 14 | 17 | 73
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 2 | 0 | 3
  Not Hispanic or Latino | 28 | 35 | 27 | 20 | 110
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 1 | 0 | 7
  White | 26 | 31 | 26 | 19 | 102
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Remission Rate Defined as the Percentage of Patients Whose Respnse is CR or CRp Based on International Working Group (IWG) Response Criteria and Treatment Outcomes Definitions
Description: Combined remission rate (complete remission [CR] + complete remission with incomplete platelet recovery [CRp]) of vosaroxin of patients ≥ 60 years old with previously untreated (de novo or secondary) AML are presented by treatment group for all treated analysis set.
  Per IWG criteria, a CR requires bone marrow blasts < 5%, absolute neutrophil count (ANC) > 1000 cells/uL, and platelet (plt) count > 100,000 plt/uL. The criteria for CRp are the same as those for CR, except for platelet count <= 100,000 lt/uL. Investigators were to determine a response category for each patient by examination of bone marrow and blood counts at the time of hematologic recovery after induction or reinduction. Investigator assessment categories included CR, CRp, CRi (Morphologic CR with incomplete blood count recovery), PR (partial remission), treatment failure, and relapse.
Time Frame: 2 years
Population: The all treated analysis set Included all enrolled patients who received any amount of vosaroxin.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Total: Schedule A, B and C combined
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4 | Total
Number analyzed (Participants) | 29 | 35 | 29 | 20 | 113
percentage of patients | 41.4 [23.5 to 61.1] | 25.7 [12.5 to 43.3] | 34.5 [17.9 to 54.3] | 25.0 [8.7 to 49.1] | 31.9 [24.3 to 41.3]

2. Secondary Outcome: Leukemia-free Survival (LFS)
Description: The censor date was the last known alive date without report of relapse.
Time Frame: 2 years
Population: All treated analysis set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4 | Total
Number analyzed (Participants) | 29 | 35 | 29 | 20 | 113
Months | 9.8 [2.4 to 15.7] | 10.9 [2.9 to 15.0] | 5.5 [1.5 to 7.3] | 4.9 [1.3 to 4.9] | 6.1 [4.9 to 9.8]

3. Secondary Outcome: Overall Survival
Time Frame: 2 years
Population: All treated patients
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Total: Schedule A, B, and C combined
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4 | Total
Number analyzed (Participants) | 29 | 35 | 29 | 20 | 113
Months | 8.6 [1.2 to 14.7] | 5.8 [1.9 to 10.1] | 7.8 [3.4 to 12.2] | 5.6 [1.8 to 11.1] | 7.0 [4.0 to 9.2]

4. Secondary Outcome: Pharmacokinetics Day 1 - Cmax (ng/mL)
Description: Pharmacokinetic Parameters (Cmax) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 1
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. The standard deviation is really CV% in the table.
Time Frame: 1 Day
Population: Patients Treated with Vosaroxin as a Single Agent (SPO-0014) on Day 1. Of 113 patients treated, PK data were available for 33 patients who received at least 1 dose of vosaroxin, PK profiles were evaluated for 10 patients in Schedule A, for 9 patients in Schedule B, for 6 patients in Schedule C, and for 8 patients in Schedule C.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 10 | 9 | 6 | 8
ng/mL | 3028 (48.7) | 2450 (47.8) | 2865 (47.8) | 3328 (69.0)

5. Secondary Outcome: Pharmacokinetics Day 4 Cmax (ng/mL)
Description: Pharmacokinetic Parameters by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) on Day 4
  Please note that N, mean and CV% are reported, but CV% is not an option in the drop down menu. So Standard Deviation is really CV% in the table.
Time Frame: Day 4
Population: Patients Treated with Vosaroxin as a Single Agent (SPO-0014) Day 4. Of 113 patients treated, PK data were available for 33 patients who received at least 1 dose of vosaroxin, PK profiles were evaluated for patients with data on Day 4 for 5 patients in Schedule C, and for 8 patients in Schedule C .
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 5 | 8
ng/mL | 5792 (114.9) | 4148 (98.4)

6. Secondary Outcome: All Cause Mortality
Description: Mortality of those patients enrolled in the study and receiving intervention
Time Frame: 30 and 60 days
Population: All treated analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4 | Total
Number analyzed (Participants) | 29 | 35 | 29 | 20 | 113
Participants
  30-Day | 5 | 3 | 2 | 2 | 12
  60-Day | 11 | 13 | 5 | 6 | 35

7. Secondary Outcome: Pharmacokinetics Day 1 - AUC0-72 and AUCinf (hr*ng/mL)
Description: Pharmacokinetic Parameters (AUC0-72 and AUCinf ) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 1
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. The standard deviation is really CV% in the table.
Time Frame: 1 Day
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 10 | 9 | 6 | 8
hr*ng/mL
  AUC0-72 (hr.ng/mL) | 36721 (21.1) | 40092 (28.7) | 37401 (13.9) | 38086 (28.0)
  AUCinf (hr.ng/mL) | 41903 (27.3) | 47228 (28.7) | 44848 (13.0) | 43838 (31.8)

8. Secondary Outcome: Pharmacokinetics Day 1 - t1/2 (hr) and MRTinf (hr)
Description: Pharmacokinetic Parameters (t1/2 and and MRTinf) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 1
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. The standard deviation is really CV% in the table.
Time Frame: 1 Day
Population: Patients Treated with Vosaroxin as a Single Agent (SPO-0014) on Day 1. Of 113 patients treated, PK data were available for 33 patients who received at least 1 dose of vosaroxin, PK profiles were evaluated for 10 patients in Schedule A, for 8 patients in Schedule B, for 6 patients in Schedule C, and for 8 patients in Schedule C.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 10 | 8 | 6 | 8
hr
  t1/2 (hr) | 22.51 (36.6) | 27.29 (21.2) | 28.27 (32.1) | 23.57 (25.2)
  MRTinf (hr) | 30.56 (41.4) | 37.57 (23.5) | 37.16 (36.8) | 32.10 (27.0)

9. Secondary Outcome: Pharmacokinetics Day 1 - CL (L/hr)
Description: Pharmacokinetic Parameters (CL) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 1
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. The standard deviation is really CV% in the table.
Time Frame: 1 Day
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 10 | 8 | 6 | 8
L/hr | 3.643 (30.0) | 3.389 (33.4) | 3.235 (15.2) | 4.538 (25.3)

10. Secondary Outcome: Pharmacokinetics Day 1 - Vss (L)
Description: Pharmacokinetic Parameters (Vss ) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 1
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. The standard deviation is really CV% in the table.
Time Frame: 1 Day
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 10 | 8 | 6 | 8
L | 107.9 (40.4) | 129.9 (50.2) | 116.6 (28.5) | 139.2 (21.1)

11. Secondary Outcome: Pharmacokinetics Day 4 - AUC0-72 and AUCinf (hr*ng/mL)
Description: Pharmacokinetic Parameters (AUC0-72 and AUCinf ) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 4
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. Standard Deviation is really CV% in the table.
Time Frame: Day 4
Population: Patients Treated with Vosaroxin as a Single Agent (SPO-0014) on Day 4. Of 113 patients treated, PK data were available for 33 patients who received at least 1 dose of vosaroxin, PK profiles were evaluated for patients with data on Day 4, for 5 patients in Schedule C, and for 8 patients in Schedule C.
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 5 | 8
hr*ng/mL
  AUC0-72 (hr.ng/mL) | 35125 (23.8) | 43667 (32.3)
  AUCinf (hr.ng/mL) | 40539 (26.9) | 46462 (37.2)

12. Secondary Outcome: Pharmacokinetics Day 4 - t1/2 (hr) and MRTinf (hr)
Description: Pharmacokinetic Parameters (t1/2 and and MRTinf) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 4
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. The Standard Deviation is really CV% in the table.
Time Frame: Day 4
Population: Patients Treated with Vosaroxin as a Single Agent (SPO-0014) on Day 4. Of 113 patients treated, PK data were available for 33 patients who received at least 1 dose of vosaroxin, PK profiles were evaluated for patients with data, for 5 patients in Schedule C, and for 7 patients in Schedule C.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 5 | 7
hr
  t1/2 (hr) | 23.52 (27.6) | 20.41 (28.7)
  MRTinf (hr) | 31.83 (35.7) | 27.79 (24.1)

13. Secondary Outcome: Pharmacokinetics Day 4 - CL (L/hr)
Description: Pharmacokinetic Parameters (CL) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 4
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. The standard deviation is really CV% in the table.
Time Frame: Day 4
Population: Patients Treated with Vosaroxin as a Single Agent (SPO-0014) on Day 4. Of 113 patients treated, PK data were available for 33 patients who received at least 1 dose of vosaroxin, PK profiles were evaluated for patients with data on Day 4, for 5 patients in Schedule C, and for 7 patients in Schedule C.
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 5 | 7
L/hr | 4.387 (30.3) | 4.882 (28.4)

14. Secondary Outcome: Pharmacokinetics Day 4 - Vss (L)
Description: Pharmacokinetic Parameters (Vss ) by Schedule, Dosing Day, and Dose Cohort for Patients Treated With Vosaroxin as a Single Agent (SPO 0014) for Day 4
  Numbers reported are N, mean and CV%. Please note CV% is not a choice that can be entered from the drop down menu. The standard deviation is really CV% in the table.
Time Frame: Day 4
Population: Patients Treated with Vosaroxin as a Single Agent (SPO-0014) on Day 4. Of 113 patients treated, PK data were available for 33 patients who received at least 1 dose of vosaroxin, PK profiles were evaluated for patients with data for Day 4, for 5 patients in Schedule C, and for 7 patients in Schedule C.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
Number analyzed (Participants) | 5 | 7
L | 137.3 (39.5) | 132.7 (34.0)

ADVERSE EVENTS:
Time Frame: Study Start: 15 May 2008, Study Completion: 23 November 2009.Treatment-Emergent Adverse Events
Arm/Group | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 | Schedule C: 72 mg/m2 on Days 1 and 4 | Schedule C: 90 mg/m2 on Days 1 and 4
All-Cause Mortality (participants affected / at risk) | 25/29 | 31/35 | 28/29 | 19/20
Serious Adverse Events (participants affected / at risk) | 25/29 | 29/35 | 21/29 | 17/20
Other Adverse Events (participants affected / at risk) | 29/29 | 35/35 | 29/29 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 (N=29) | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 (N=35) | Schedule C: 72 mg/m2 on Days 1 and 4 (N=29) | Schedule C: 90 mg/m2 on Days 1 and 4 (N=20)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 6 | 6 | 6
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 1 | 0
Cardio-Respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Intestinal functional disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 3 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0 | 0
Multi-Organ failure (General disorders) | 1 | 0 | 0 | 0
Non-Cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 2 | 3 | 2 | 2
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis orbital (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 5 | 11 | 7 | 4
Pneumonia fungal (Infections and infestations) | 1 | 0 | 1 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 3 | 2 | 2
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis fungal (Infections and infestations) | 0 | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1 | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Streptococcal bacteraemia (Infections and infestations) | 1 | 0 | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Ejection fraction decreased (Investigations) | 0 | 0 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 1 | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Schedule A: 72 mg/m2 Vosaroxin Days 1, 8 and 15 (N=29) | Schedule B: 72 mg/m2 Vosaroxin on Days 1 and 8 (N=35) | Schedule C: 72 mg/m2 on Days 1 and 4 (N=29) | Schedule C: 90 mg/m2 on Days 1 and 4 (N=20)
Anaemia (Blood and lymphatic system disorders) | 12 | 19 | 19 | 12
Coagulopathy (Blood and lymphatic system disorders) | 1 | 4 | 2 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 10 | 19 | 14 | 5
Hilar lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 5 | 0 | 1
Lymph node calcification (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 9 | 8 | 5
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Splenomegaly (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 12 | 24 | 20 | 12
Acute myocardial infraction (Cardiac disorders) | 0 | 1 | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 1 | 4 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 4 | 4 | 6 | 4
Atrial flutter (Cardiac disorders) | 0 | 1 | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 0 | 2 | 3
Bundle branch block (Cardiac disorders) | 0 | 1 | 0 | 0
Bundle branch block left (Cardiac disorders) | 1 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 2 | 1 | 2 | 0
Cardiomegaly (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0
Left ventricular failure (Cardiac disorders) | 0 | 0 | 2 | 0
Mitral valve Disease (Cardiac disorders) | 0 | 1 | 0 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infraction (Cardiac disorders) | 1 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 2 | 0
Pericardial cyst (Cardiac disorders) | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 1 | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 1 | 5 | 3 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 11 | 14 | 5 | 5
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 0 | 1 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 1 | 1 | 1
Spondylolisthesis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1
Cerumen impaction (Ear and labyrinth disorders) | 0 | 1 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 2 | 0 | 1 | 0
Eustachian tube patulous (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 1 | 0 | 0
Conjunctival discolouration (Eye disorders) | 0 | 0 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 0
Dry eye (Eye disorders) | 1 | 1 | 1 | 0
Erythema of eyelid (Eye disorders) | 1 | 1 | 0 | 0
Eye haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Eye Oedema (Eye disorders) | 0 | 1 | 0 | 0
Eye Pruritus (Eye disorders) | 0 | 0 | 0 | 1
Eyelid disorder (Eye disorders) | 0 | 0 | 1 | 0
Eyelid oedema (Eye disorders) | 0 | 1 | 0 | 0
Eyelid ptosis (Eye disorders) | 0 | 1 | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0
Madarosis (Eye disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Ocular icterus (Eye disorders) | 1 | 1 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 3 | 0 | 0 | 1
Visual disturbance (Eye disorders) | 1 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 1 | 1 | 0
Vitreous floaters (Eye disorders) | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 5 | 5 | 6
Abdominal pain (Gastrointestinal disorders) | 9 | 6 | 6 | 3
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 5 | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Anorectal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Aptyalism (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Bowel sounds abnormal (Gastrointestinal disorders) | 1 | 3 | 0 | 1
Breath odour (Gastrointestinal disorders) | 2 | 1 | 0 | 0
Caecitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 1 | 3 | 0 | 0
Colonic Pseudo-obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 12 | 13 | 5 | 4
Dental discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 24 | 27 | 20 | 14
Diverticulum (Gastrointestinal disorders) | 2 | 1 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 6 | 5 | 4 | 3
Dyspepsia (Gastrointestinal disorders) | 5 | 3 | 6 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 9 | 6 | 1
Enlarged uvula (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Faecal incontinence (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 3 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 5 | 0 | 1
Gingival swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gingivitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 5 | 7 | 2 | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Leukoplakia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip blister (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip dry (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Lip haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Lip ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Malabsorption (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 1 | 3 | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 22 | 21 | 25 | 11
Odynophagia (Gastrointestinal disorders) | 4 | 1 | 0 | 1
Oedema mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal disorder (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal Spasm (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Oral discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral mucosal blistering (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral mucosal discolouration (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Oral mucosal petechiae (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 2 | 5 | 5 | 6
Oral soft tissue disorder (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Palatal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Perianal erythema (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Poor dental condition (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 1 | 3 | 1
Rectal fissure (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Rectal spasm (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Salivary gland disorder (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 18 | 19 | 15 | 11
Tongue blistering (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue discolouration (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Tongue haematoma (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Tongue haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tongue oedema (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 16 | 10 | 15 | 6
Application site hypersensitivity (General disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 9 | 14 | 6 | 3
Axillary pain (General disorders) | 0 | 0 | 1 | 0
Catheter related complication (General disorders) | 2 | 1 | 3 | 2
Catheter site erythema (General disorders) | 1 | 3 | 1 | 2
Catheter site excoriation (General disorders) | 1 | 0 | 0 | 0
Catheter site haematoma (General disorders) | 0 | 0 | 1 | 0
Catheter site haemorrhage (General disorders) | 1 | 1 | 0 | 0
Catheter site inflammation (General disorders) | 1 | 0 | 0 | 0
Catheter site oedema (General disorders) | 1 | 0 | 0 | 0
Catheter site pain (General disorders) | 1 | 3 | 5 | 1
Catheter site related reaction (General disorders) | 0 | 0 | 2 | 0
Catheter Thrombosis (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 1 | 0
Chest pain (General disorders) | 3 | 3 | 4 | 1
Chills (General disorders) | 8 | 12 | 8 | 6
Discomfort (General disorders) | 0 | 0 | 1 | 0
Early Satiety (General disorders) | 0 | 0 | 0 | 1
Face Oedema (General disorders) | 0 | 1 | 0 | 0
Facial pain (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 15 | 20 | 12 | 7
Feeling cold (General disorders) | 1 | 0 | 1 | 0
Gait disturbance (General disorders) | 1 | 2 | 0 | 0
Generalized oedema (General disorders) | 1 | 4 | 1 | 1
Induration (General disorders) | 0 | 0 | 2 | 0
Infusion site pain (General disorders) | 1 | 0 | 0 | 0
Injection site bruising (General disorders) | 1 | 0 | 0 | 0
Injection site reaction (General disorders) | 1 | 0 | 1 | 0
Malaise (General disorders) | 6 | 2 | 2 | 2
Mucosal Inflammation (General disorders) | 1 | 2 | 0 | 0
Mucous membrane disorder (General disorders) | 0 | 0 | 0 | 1
Multi-Organ failure (General disorders) | 0 | 1 | 0 | 0
Nodule (General disorders) | 1 | 0 | 0 | 0
Non-Cardiac chest pain (General disorders) | 1 | 1 | 2 | 1
Oedema (General disorders) | 2 | 1 | 0 | 1
Oedema peripheral (General disorders) | 17 | 17 | 15 | 9
Pain (General disorders) | 5 | 2 | 7 | 3
Performance status decreased (General disorders) | 0 | 1 | 0 | 0
Peripheral coldness (General disorders) | 0 | 1 | 2 | 0
Pyrexia (General disorders) | 5 | 9 | 7 | 7
Suprapubic pain (General disorders) | 0 | 0 | 0 | 1
Swelling (General disorders) | 1 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1 | 0 | 0
Abscess (Infections and infestations) | 1 | 0 | 0 | 0
Acinetobacter bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Anorectal infection bacterial (Infections and infestations) | 0 | 1 | 2 | 0
Bacteraemia (Infections and infestations) | 2 | 3 | 0 | 1
Bacterial infection (Infections and infestations) | 1 | 1 | 0 | 0
Bacteroides bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Candidiasis (Infections and infestations) | 3 | 4 | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 1 | 0 | 0
Catheter site cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 1 | 0
Central line infection (Infections and infestations) | 0 | 1 | 0 | 0
Chronic Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridial infection (Infections and infestations) | 0 | 1 | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 2 | 0 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 3 | 3 | 0 | 1
Enterococcal infection (Infections and infestations) | 2 | 0 | 1 | 1
Epiglottitis (Infections and infestations) | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 2 | 1
Fungaemia (Infections and infestations) | 1 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 2 | 0
Fungal rash (Infections and infestations) | 0 | 0 | 1 | 0
Fusarium infection (Infections and infestations) | 1 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 1 | 0 | 0
Herpes simplex (Infections and infestations) | 2 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Localized infection (Infections and infestations) | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0
Oral Candidiasis (Infections and infestations) | 0 | 1 | 1 | 2
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 3 | 4 | 3
Pneumonia fungal (Infections and infestations) | 1 | 1 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 1 | 0
Rectal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 1 | 2 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 3 | 3 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 0 | 0
Stenotrophomonas infection (Infections and infestations) | 0 | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1 | 0 | 2
Urinary tract infection enterococcal (Infections and infestations) | 2 | 0 | 0 | 1
Urinary tract infection fungal (Infections and infestations) | 0 | 0 | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 1 | 0 | 1
Urinary tract infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0
Vaginal candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Anaphylactic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 2 | 2 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 3 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Incision site erythema (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 5 | 3 | 1
Skin injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 3 | 2 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tracheal deviation (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 3 | 1 | 3 | 2
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 2 | 2 | 2 | 0
Wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 0 | 0
Bacteria sputum identified (Investigations) | 0 | 2 | 0 | 0
Bacteria urine identified (Investigations) | 1 | 0 | 0 | 0
Bacterial culture positive (Investigations) | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 3 | 3 | 0 | 1
Blood culture positive (Investigations) | 0 | 0 | 1 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0
Blood testosterone decreased (Investigations) | 1 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 0 | 1 | 0
Body temperature decreased (Investigations) | 1 | 0 | 0 | 0
Breath sounds abnormal (Investigations) | 7 | 6 | 3 | 1
C-Reactive protein increased (Investigations) | 1 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 4 | 0 | 0
Chest x-ray abnormal (Investigations) | 1 | 2 | 1 | 0
Clostridium difficile toxin test positive (Investigations) | 0 | 0 | 0 | 1
Culture urine positive (Investigations) | 0 | 0 | 1 | 0
Ejection fraction decreased (Investigations) | 2 | 0 | 1 | 0
Electrocardiogram qrs complex abnormal (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram qt corrected interval prolonged (Investigations) | 0 | 0 | 1 | 1
Electrocardiogram qt prolonged (Investigations) | 0 | 1 | 0 | 0
Electrocardiogram st segment abnormal (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram st segment depression (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram st-t change (Investigations) | 1 | 1 | 0 | 0
Electrocardiogram st-t segment abnormal (Investigations) | 0 | 0 | 0 | 1
Electrocardiogram t wave abnormal (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram t wave inversion (Investigations) | 1 | 0 | 0 | 0
Heart rate irregular (Investigations) | 1 | 0 | 1 | 0
Helicobacter pylori identification test positive (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 1
Hepatitis a antibody positive (Investigations) | 0 | 1 | 0 | 0
International normalised ratio increased (Investigations) | 4 | 2 | 2 | 3
Liver function test abnormal (Investigations) | 0 | 1 | 1 | 0
Liver scan abnormal (Investigations) | 0 | 1 | 0 | 0
Lymph node palpable (Investigations) | 1 | 1 | 0 | 0
Nuclear magnetic resonance imaging brain abnormal (Investigations) | 0 | 1 | 0 | 0
Oxygen consumption increased (Investigations) | 0 | 1 | 0 | 0
Oxygen saturation decreased (Investigations) | 0 | 2 | 1 | 0
Prostate examination abnormal (Investigations) | 0 | 0 | 2 | 0
Prothrombin level increased (Investigations) | 1 | 0 | 0 | 0
Prothrombin time prolonged (Investigations) | 1 | 0 | 0 | 0
Pulse pressure decreased (Investigations) | 0 | 2 | 1 | 0
Pulse pressure increased (Investigations) | 0 | 1 | 0 | 0
Radial pulse abnormal (Investigations) | 0 | 2 | 0 | 0
Respiratory rate increased (Investigations) | 0 | 0 | 1 | 0
Skin turgor decreased (Investigations) | 1 | 4 | 0 | 1
Sputum culture positive (Investigations) | 0 | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 2 | 0 | 0
Troponin i increased (Investigations) | 0 | 0 | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1 | 0 | 0
Urine colour abnormal (Investigations) | 0 | 2 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0 | 1
Weight decreased (Investigations) | 6 | 3 | 3 | 3
Weight increased (Investigations) | 0 | 0 | 1 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0 | 0
X-Ray abnormal (Investigations) | 0 | 1 | 0 | 0
Xanthochromia (Investigations) | 0 | 1 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 21 | 18 | 17 | 11
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 4 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 7 | 3 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Diabetes mellitus insulin-dependent (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 2 | 3 | 4 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 7 | 6 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 3 | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 4 | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 5 | 9 | 4
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 21 | 19 | 17 | 14
Hypomagnesaemia (Metabolism and nutrition disorders) | 15 | 14 | 14 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 6 | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 8 | 6 | 6
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 3 | 2 | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Oral intake reduced (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5 | 4 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 7 | 5 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 4 | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 3 | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 4 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4 | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 5 | 7 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Spondylolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Ageusia (Nervous system disorders) | 0 | 1 | 0 | 0
Aphasia (Nervous system disorders) | 0 | 1 | 0 | 0
Carotid artery occlusion (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0
Coordination abnormal (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 6 | 7 | 7 | 4
Dysarthria (Nervous system disorders) | 2 | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 5 | 3 | 5
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Extrapyramidal disorder (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 10 | 9 | 9 | 2
Hemiparesis (Nervous system disorders) | 0 | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 1
Hypogeusia (Nervous system disorders) | 1 | 0 | 2 | 0
Hyporeflexia (Nervous system disorders) | 0 | 1 | 0 | 0
Hyposmia (Nervous system disorders) | 0 | 0 | 1 | 0
Intention tremor (Nervous system disorders) | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 1 | 2 | 4 | 3
Memory impairment (Nervous system disorders) | 0 | 0 | 1 | 0
Nervous system disorder (Nervous system disorders) | 0 | 1 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 2 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Parosmia (Nervous system disorders) | 0 | 0 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0
Periventricular leukomalacia (Nervous system disorders) | 0 | 1 | 0 | 0
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 4 | 4 | 2 | 1
Speech disorder (Nervous system disorders) | 0 | 2 | 0 | 0
Syncope (Nervous system disorders) | 0 | 2 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0 | 0
Tremor (Nervous system disorders) | 1 | 2 | 2 | 0
Agitation (Psychiatric disorders) | 6 | 0 | 4 | 3
Anxiety (Psychiatric disorders) | 7 | 14 | 12 | 4
Apathy (Psychiatric disorders) | 0 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 8 | 9 | 7 | 3
Delirium (Psychiatric disorders) | 2 | 0 | 0 | 0
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 5 | 5 | 6 | 2
Disorientation (Psychiatric disorders) | 0 | 1 | 1 | 0
Dysthymic disorder (Psychiatric disorders) | 0 | 1 | 0 | 0
Flat affect (Psychiatric disorders) | 0 | 1 | 0 | 0
Hallucination (Psychiatric disorders) | 2 | 1 | 0 | 2
Insomnia (Psychiatric disorders) | 12 | 13 | 11 | 3
Mental disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 3 | 2 | 1
Mood altered (Psychiatric disorders) | 0 | 1 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 1 | 0
Restlessness (Psychiatric disorders) | 3 | 3 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1 | 0
Bladder diverticulum (Renal and urinary disorders) | 0 | 0 | 1 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 3 | 0 | 1 | 0
Haematuria (Renal and urinary disorders) | 4 | 11 | 2 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 2 | 3 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 2 | 0
Nocturia (Renal and urinary disorders) | 1 | 1 | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 2 | 2
Renal cyst (Renal and urinary disorders) | 1 | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 3 | 2 | 0
Renal mass (Renal and urinary disorders) | 1 | 0 | 0 | 0
Residual urine (Renal and urinary disorders) | 1 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 3 | 4 | 1 | 2
Urinary retention (Renal and urinary disorders) | 2 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic fluid collection (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Penile oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Penile pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Scrotal erythema (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vulval disorder (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 13 | 11 | 11 | 6
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 11 | 6
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1
Epiglottic oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 13 | 8 | 5
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 6 | 2
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pharyngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 4 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 11 | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 1
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 4 | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 10 | 8 | 2 | 4
Respiratory alkalosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 6 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0 | 0
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 3
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 8 | 13 | 5
Blister (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 5 | 3 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 8 | 7 | 4 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 3 | 8 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 5 | 5 | 2
Leukocytoclastic vasculitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 2 | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Penile ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Perivascular dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 8 | 11 | 4 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 5 | 6 | 1
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 7 | 8 | 9 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Red man syndrome (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Scab (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 3 | 2 | 1 | 1
Skin nodule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Sinus operation (Surgical and medical procedures) | 1 | 0 | 0 | 0
Aortic arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0
Arterial disorder (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 2 | 0 | 0
Flushing (Vascular disorders) | 1 | 2 | 2 | 0
Haematoma (Vascular disorders) | 2 | 2 | 4 | 1
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 2 | 0
Hypertension (Vascular disorders) | 6 | 4 | 3 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 11 | 11 | 10 | 6
Orthostatic hypotension (Vascular disorders) | 1 | 1 | 2 | 0
Pallor (Vascular disorders) | 4 | 3 | 2 | 0
Phlebitis (Vascular disorders) | 0 | 1 | 0 | 1
Raynaud's phenomenon (Vascular disorders) | 0 | 0 | 0 | 1
Thrombophlebitis superficial (Vascular disorders) | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 1 | 1
Bacteria tissue specimen identified (Investigations) | 0 | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 1 | 0 | 2

LIMITATIONS AND CAVEATS:
Due to the limited sample size in this study, further study is needed to confirm these results. No statistical testings were performed to compare any of the treatment groups. No p-values or odds ratios were reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days